CLINICAL TRIAL: NCT05070026
Title: Comparison of Inflammatory Cytokine Levels Between Single-port and Three-port Thoracoscopic Lobectomy in the Treatment of Non-small Cell Lung Cancer
Brief Title: Comparison of Inflammatory Cytokine Levels Between Single-port and Three-port Thoracoscopic Lobectomy in the Treatment of Non-small Cell Lung Cancersurgery on Perioperative Clinical Indexes、Inflammatory Reaction and Quality of Life Scores of Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, principal investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: uni-portal and three port VATS
Record Dates: First submitted 2021-09-12; First posted 2021-10-06 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Video-assisted Thoracoscopic Surgery; Inflammatory Reaction; Life Scores
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- uni-portal VATS group (Experimental)
  Interventions: Other: uni-portal VATS group
- three port VATS group (Experimental)
  Interventions: Other: three port VATS group

INTERVENTIONS:
Other: uni-portal VATS group — patients received pulmonary lobectomy under general anesthesia by using uni-portal VATS method
  Arms: uni-portal VATS group
Other: three port VATS group — patients received pulmonary lobectomy under under general anesthesia by using three port VATS method
  Arms: three port VATS group

SUMMARY:
Many recent studies have shown that surgical trauma will result in an immunosuppressive state. Combined with the effect of surgical stress, it will often lead to metabolic changes, systemic inflammatory response, and other problems. The body resists and removes the harmful factors through the inflammatory reaction. However, an excessive reaction will damage the normal tissues and cells of the body. The smooth recovery of the body needs to balance the degree of inflammatory reaction. Surgical patients will trigger different degrees of an inflammatory response due to different degrees of physical trauma, which runs through the process of postoperative recovery from the beginning of surgery and often prolongs the time of postoperative recovery. Reducing the intraoperative and postoperative inflammatory response of patients has always been the goal of surgeons, and a method is the reduction of surgical trauma.

The successful experience of the first single-port thoracoscopic wedge resection of the lung in 2004 provided us with a new surgical idea. Subsequently, a large number of domestic and international studies and case reports show that single-port thoracoscopic surgery is safe and feasible in lobectomy and segmental resection. With the rapid development of single-port thoracoscopic surgery in recent years, the scope of application and clinical efficacy of the surgery are gradually becoming equivalent to the traditional three-port thoracoscopic surgery, which can ensure the safety of the operation and complete tumor resection, and has its own characteristics and advantages compared with the traditional three-port thoracoscopic surgery. The reduction of incisions can significantly improve the postoperative pain and recovery of patients and wound healing.

In addition, single-port thoracoscopic surgery also has a subtle improvement in patients' intraoperative and postoperative inflammatory response compared with traditional three-port thoracoscopic surgery. In this study, we compared and analyzed the intraoperative and postoperative inflammatory factor levels of single-port thoracoscopic surgery and three-port thoracoscopic surgery in patients with non-small cell lung cancer (NSCLC). Through the comparison of the measured values, we further discussed the advantages of single-port thoracoscopic surgery in reducing inflammatory response and its application and promotion value in the treatment of patients with NSCLC compared with traditional three-port thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* (1) NSCLC was diagnosed by imaging examination (chest enhanced computed tomography or positron emission tomography-computed tomography) and biopsy pathology; (2) TNM stage was stage I and II; (3) the patient had indications of radical operation; (4) the patient had good cardiopulmonary, liver, and kidney function and no obvious surgical contraindication before operation; (5) the preoperative inflammatory indexes of all patients were within the normal range

Exclusion Criteria:

* (1) the thoracoscopic operation was converted to thoractomy; (2) the operation time was more than 3 hours; (3) blood vessel rupture occurred during the operation, and the bleeding amount was more than 200 mL; (4) the patient had complications (the patient had fever exceeding 38.5 ℃, chest computed tomography confirmed intrapulmonary infection, incision infection, postoperative bleeding, requiring secondary thoracotomy, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
intraoperative hemorrhage volume | at the end of the surgery
  record intraoperative hemorrhage volume at the end of the surgery
chest drainage time | before remove drainage tube
  record chest drainage time until remove drainage tube
duration of the healing of incision | before suture removal
  record the duration of the healing of incision
out-of-bed activity time (Day) and length of hospital stay (Day) | Before discharge from hospital
  record the days of patients' out-of-bed activity time and length of hospital stay after surgery
postoperative pain | 24 hours after surgery
  record postoperative pain 24 hours after surgery by using visual analog scale (VAS) score, where 0 indicates painlessness, and 10 indicates severe pain
postoperative adverse effects | 24 hours after surgery
  record postoperative adverse effects 24 hours after surgery
preoperative inflammation | two days before operation
  record c-reactive protein after surgery
inflammation at end of operation | end of operation
  record c-reactive protein after surgery
postoperative inflammation | 30mins after operation
  record c-reactive protein after surgery
postoperative inflammation | Day 1 after operation
  record c-reactive protein after surgery
postoperative inflammation | Day 3 after operation
  record c-reactive protein after surgery
preoperative inflammation | two days before operation
  record serum amyloid A protein (SAA) after surgery
inflammation at end of operation | end of operation
  record serum amyloid A protein (SAA) after surgery
postoperative inflammation | 30mins after operation
  record serum amyloid A protein (SAA) after surgery
postoperative inflammation | Day 1 after operation
  record serum amyloid A protein (SAA) after surgery
postoperative inflammation | Day 3 after operation
  record serum amyloid A protein (SAA) after surgery
preoperative inflammation | two days before operation
  record IL-6 after surgery
inflammation at end of operation | end of operation
  record IL-6 after surgery
postoperative inflammation | 30mins after operation
  record IL-6 after surgery
postoperative inflammation | Day 1 after operation
  record IL-6 after surgery
postoperative inflammation | Day 7 after operation
  record IL-6 after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China